CLINICAL TRIAL: NCT02289183
Title: Prospective Randomized Controlled Trial on Clinical Application Value of Modified Delta-shaped Gastroduodenostomy in Totally Laparoscopic Surgery and Billroth-I Anastomosis in Laparoscopy-assisted Surgery for Distal Gastric Cancer
Brief Title: Prospective Study on Modified Delta-shaped Gastroduodenostomy in Totally Laparoscopic Surgery for Distal Gastric Cancer
Acronym: MDSG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Fujian Medical University Union Hospital, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-01
Record Dates: First submitted 2014-11-04; First posted 2014-11-13 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Stomach Neoplasms
Keywords: Stomach Neoplasms; Laparoscopy; Billroth I Operation
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Totally laparoscopic distal gastrectomy (Experimental): The totally laparoscopic distal gastrectomy with modified delta-shaped gastroduodenostomy will be performed for the treatment of patients with distal gastric cancer assigned to this group.
  Interventions: Procedure: Totally laparoscopic distal gastrectomy
- Laparoscopy-assisted distal gastrectomy (Active Comparator): The laparoscopy-assisted distal gastrectomy with Billroth-I anastomosis will be performed for the treatment of patients with distal gastric cancer assigned to this group.
  Interventions: Procedure: Laparoscopy-assisted distal gastrectomy

INTERVENTIONS:
Procedure: Totally laparoscopic distal gastrectomy — Totally laparoscopic distal gastrectomy with modified delta-shaped gastroduodenostomy
  Arms: Totally laparoscopic distal gastrectomy
Procedure: Laparoscopy-assisted distal gastrectomy — Laparoscopy-assisted distal gastrectomy with Billroth-I anastomosis
  Arms: Laparoscopy-assisted distal gastrectomy

SUMMARY:
The purpose of this study is to explore the clinical application value of modified delta-shaped gastroduodenostomy in totally laparoscopic surgery for distal gastric cancer.

DETAILED DESCRIPTION:
A prospective randomized comparison of the modified delta-shaped gastroduodenostomy in totally laparoscopic surgery and Billroth-I anastomosis in laparoscopy-assisted surgery for distal gastric cancer will be performed, to evaluate the clinical value and provide theoretical basis and clinical experience for the extensive application of the modified technique. The evaluation parameters are perioperative clinical efficacy, postoperative life quality, immune function and 3-year survival and recurrence rates.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 75 years (including 18 and 75 years old)
* Primary distal gastric adenocarcinoma (papillary, tubular, mucinous, signet ring cell, or poorly differentiated) confirmed pathologically by endoscopic biopsy
* cT1-4a, N0-3, M0 at preoperative evaluation according to the American Joint Committee on Cancer (AJCC) Cancer Staging Manual Seventh Edition
* Expected curative resection through distal subtotal gastrectomy with D2 lymphadenectomy
* Performance status of 0 or 1 on Eastern Cooperative Oncology Group scale (ECOG)
* American Society of Anesthesiology score (ASA) class I, II, or III
* Written informed consent

Exclusion Criteria:

* Women during pregnancy or breast-feeding
* Severe mental disorder
* History of previous upper abdominal surgery (except laparoscopic cholecystectomy)
* History of previous gastrectomy, endoscopic mucosal resection or endoscopic submucosal dissection
* Enlarged or bulky regional lymph node diameter over 3cm by preoperative imaging
* History of other malignant disease within past five years
* History of previous neoadjuvant chemotherapy or radiotherapy
* History of unstable angina or myocardial infarction within past six months
* History of cerebrovascular accident within past six months
* History of continuous systematic administration of corticosteroids within one month
* Requirement of simultaneous surgery for other disease
* Emergency surgery due to complication (bleeding, obstruction or perforation) caused by gastric cancer
* FEV1<50% of predicted values

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival rate | 36 months

SECONDARY OUTCOMES:
Morbidity and mortality | 30 days;36 months
  The early postoperative complication and mortality are defined as the event observed within 30 days after surgery, while the time frame for late complication is the period from postoperative day 31th to the end of month 36th.
Intraoperative situation | 1 day
  Operation time, intraoperative blood loss and transfusion volume, conversive rate, intraoperative bleeding and viscera damage, and incision length are used to access the intraoperative situation
Postoperative recovery course | 10 days
  Time to first ambulation, flatus, liquid diet and soft diet, duration of postoperative hospital stay and postoperative pain are used to assess the postoperative recovery course.Visual analog pain score method is used to evaluate the difference of postoperative pain degree.
Postoperative nutritional status and quality of life | 12 months
  The variation of weight, cholesterol and albumin on postoperative 3, 6, 9 and 12 months, and the results of endoscopy on postoperative 3 and 12 months are used to access the postoperative nutritional status and quality of life.
Inflammatory and immune response | 7 days
  The daily highest body temperature before discharge and the values of white blood cell count, hemoglobin, C-reactive protein, prealbumin and relevant immune cytokines including T cell percentage, T-helper lymphocytes (CD4+) percentage, T-suppressor lymphocytes (CD8+) percentage, natural killer (NK) cells percentage from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded.
3-year overall survival rate | 36 months
3-year recurrence pattern | 36 months
  Recurrence patterns are classified into five categories at the time of first diagnosis: locoregional, hematogenous, peritoneal, distant lymph node, and mixed type.

CONTACTS AND LOCATIONS:
Overall Officials: Changming Huang, M.D.,Ph.D., Study Chair — Fujian Medical University Union Hospital; Chaohui Zheng, M.D., Study Director — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No